CLINICAL TRIAL: NCT04395469
Title: Feasibility Study of Hypoxia and Re-oxygenation Imaging in Pancreatic Cancer Using Positron Emission Tomography (PET) With [18F] Fluoroazomycin-arabinoside (FAZA PET) and Magnetic Resonance Imaging (MRI)
Brief Title: FAZA PET/MRI Pancreas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 19-6358-C
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Adenocarcinoma Non-resectable; Locally Advanced Pancreatic Adenocarcinoma; Unresectable Pancreatic Cancer
Keywords: Hypoxia; FAZA; PET Imaging; FAZA PET MRI; locally advanced un-resectable pancreatic adenocarcinoma; Unresectable; Non-metastatic
MeSH Terms: conditions — Hypoxia | interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: 18F-FAZA — 18F-FAZA is a radiotracer used for PET imaging (in combination with MRI) to detect hypoxia in tumours. This scan will be done before and after radiation treatment.

SUMMARY:
This is a single arm, single centre, investigator initiated study to investigate the use of FAZA-PET in combination with MRI. FAZA is an investigational radiotracer used in PET scans. FAZA PET-MRI will be used to measure hypoxia in up to 20 patients with unresectable, non-metastatic, locally advanced un-resectable pancreatic adenocarcinoma (LAPAC).

After each FAZA PET-MRI scan, patients will be followed up via telephone, 48 hours after the imaging session to assure that the procedure was tolerated without side effects. Patients will undergo a FAZA PET-MRI scans before and after their standard of care radiation treatment.

DETAILED DESCRIPTION:
The success of hypoxia-targeted therapies has so far been limited, a fact widely attributed to the absence of a reliable imaging biomarker for hypoxia that could easily be implemented into a routine clinical workflow. A compelling study has found the presence of hypoxia in pancreatic tumors using FAZA-PET imaging. The data derived from this alternative dual-imaging approach can be used to establish a patient-specific perfusion-to-hypoxia mapping, accounting for differences in tumour metabolisms. This technique was recently validated in a pre-clinical FAZA-PET/CE-MRI study of mice with orthotopically-implanted pancreatic patient-derived tumour xenografts.

The purpose of this study is to look for hypoxia in tumours using a PET scan in combination with MRI. The use of PET/MRI scans to measure hypoxia may be better and simpler than the approaches used previously. This study will assess whether or not PET/MRI scans can provide useful information about hypoxia in pancreatic cancer. Additionally, a recent study at the Princess Margaret Cancer Centre found varying levels of hypoxia in patients with pancreatic tumors, providing a rationale for incorporating hypoxia imaging and patient-specific treatment adaptation into the clinical management of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. One or more of the following:

   A) Participants who have histologically confirmed new diagnosis of unresectable, non-metastatic, LAPAC as assessed by the multidisciplinary tumor board based on pre-RT imaging and clinical assessment, and are amenable to SBRT.

   B) Patients who received prior systemic therapy for unresectable LAPAC may be consented and enrolled if they still have localized unresectable LAPAC amenable to SBRT.

   C) Participants with newly diagnosed LAPAC who received systemic therapy for borderline resectable pancreatic adenocarcinoma and have become unresectable following preoperative multidisciplinary assessment, are eligible for the study if the patient meets the eligibility criteria based on staging following systemic therapy.

   D) Participants with newly diagnosed borderline resectable pancreatic adenocarcinoma.
2. Age ≥18 years.
3. ECOG performance status ≤2 (see Appendix A).
4. Life expectancy of greater than 6 months.
5. A negative serum pregnancy test prior to PET-MR imaging, for women of child-bearing age.
6. Ability to understand and the willingness to sign a written informed consent document.
7. Eligible for treatment on the integrated magnet resonance linear accelerator (MRL).

Exclusion Criteria:

1. Patients who have had prior RT to upper abdomen.
2. Patients who are receiving any other concomitant investigational agents. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
3. Patients with early stage resectable (I-II) pancreatic cancer, or known distant metastases.
4. Contraindication to MRI scan as per current institutional guidelines.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Pregnant women are excluded from this study because of the potential teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants, breastfeeding should be discontinued.
7. Patients who have a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin (other than head and neck region), or carcinoma in situ (e.g., in situ cervical cancer or breast carcinoma) that have undergone potentially curative therapy are not excluded.
8. History or current evidence of any condition, therapy, or laboratory abnormality, known psychiatric or substance abuse disorders that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Tumor Hypoxia | 2.5 years
  Hypoxic regions in the tumour are defined as regions for which the voxel-scale activity exceeds the mean activity in the left-ventricle blood pool by a ratio of 1.2. The fraction of such voxels in a given tumour defines the hypoxic fraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada